CLINICAL TRIAL: NCT00745966
Title: A 8-Week, Multicenter, Open-Label, Observational Study of Atypical Antipsychotics in Improvement of Quality of Life in Bipolar Disorder
Brief Title: Atypical Antipsychotics in Improvement of Quality of Life in Bipolar Disorder
Acronym: POLE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Joon-Woo Bahn, AstraZeneca
Other Study IDs: NIS-NKR-SER-2008/1
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-09

CONDITIONS: Naturalistic; Observational
Keywords: Bipolar; atypical antipsychotics; quality of life; observational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to reassure the clinical study data on atypical antipsychotics effect on quality of life in Korean Bipolar patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient and the patient's legal representative (if any) must understand the nature of the study and must have given written consent.
* Meet DSM-IV-TR criteria for bipolar disorder (bipolar I disorder, bipolar II disorder) at the time of baseline.

Exclusion Criteria:

* Serious or unstable, medical illness. Subjects with chronic illness may be included but must be stable and otherwise physically healthy on the basis of a physical examination, medical history.
* Known intolerance for or lack of response to atypical antipsychotics , as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The change from the baseline to week 8 in Short Form of the Quality of Life Enjoyment and satisfaction Questionnaire (Q-LES-Q) score

SECONDARY OUTCOMES:
The change from the baseline to week 8 in CGI-BP and GAF scale score.

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Woo Bahn, Study Director — Astrazeneca, Korea
Locations (2):
- South Korea (2):
  - Research Site, Kyunggi-do, Choonchun-si
  - RFesearch Site, Daegu, Joong-gu